CLINICAL TRIAL: NCT05803811
Title: Effect of Colon Delivered Vitamin B2 on Gut Microbiota and Related Health Biomarkers in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-11-11-VITB2
Record Dates: First submitted 2023-02-16; First posted 2023-04-07 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-09

CONDITIONS: Quality of Life
Keywords: microbiota; vitaminB2; Riboflavin; ShortChain fatty acids
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose (Experimental): Daily dose of 1.4 mg of Vitamin B2 (Riboflavin) once a day for 12 weeks
  Interventions: Dietary Supplement: Riboflavin
- Mid dose (Experimental): Daily dose of 10 mg of Vitamin B2 (Riboflavin) once a day for 12 weeks
  Interventions: Dietary Supplement: Riboflavin
- high dose (Experimental): Daily dose of 75 mg Vitamin B2 (Riboflavin) once a day for 12 weeks
  Interventions: Dietary Supplement: Riboflavin
- Placebo (Placebo Comparator): One capsule of 570 mg (consisting of microcrystalline cellulose) once a day for 12 weeks
  Interventions: Dietary Supplement: Riboflavin

INTERVENTIONS:
Dietary Supplement: Riboflavin — Colon delivered vitamin B2 (Riboflavin) for 12 weeks

SUMMARY:
The goal of this intervention study (clinical trial) is to investigate the effect of colon-delivered Riboflavin (vitamin B2) on the faecal microbial composition and diversity in older healthy subjects (50 -70 years of age)

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be willing and able to give written informed consent and to understand, to participate, and to comply with the clinical study requirements.
2. Between 50 and 70 years of age.
3. Has a BMI of between 18.5 - 30 Kg/m2.
4. Participants have had a stable body weight (≤5 % change) over the past 3-months.
5. Is in general good health, as determined by interview and vital signs (blood pressure, heart rate, pulse) by the investigator.
6. Willing to avoid consuming gut microbiome modulating dietary supplements, prebiotic, probiotic, or fibre-rich supplements, and, within 4 weeks prior to the baseline visit, until the end of the study.
7. Maintain current level of physical activity.
8. Willing to consume the investigational product daily for the duration of the study.
9. Female participants in menopause for at least the last one year. -

Exclusion Criteria:

1. Are hypersensitive to any of the components of the test product.
2. Has taken antibiotics within the previous 3 months prior to Baseline (Visit2)
3. Is currently using systemic steroids, systemic antibiotics, proton pump inhibitors, H2 blocker, antacid, metformin, or immunosuppressant medication.
4. Participant has a history of drug and/or alcohol abuse at the time of enrolment (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); Is currently in treatment for alcohol/substance abuse; Has been diagnosed with alcohol/substance abuse disorder).
5. Is a smoker or vaper.
6. Vegetarian or vegan.
7. Has made any major dietary changes in the past 3 months prior to Baseline (Visit 2).
8. Planned major changes in the lifestyle (i.e., diet, dieting, exercise level, significant travel) during the duration of the study.
9. Has a currently active eating disorder.
10. Has food allergies or other issues with foods that would preclude the intake of the study products, as determined by the study investigator.
11. Is having a typical fibre intake >30 g fibre/day.
12. Has an active gastrointestinal disorder or previous gastrointestinal surgery, which in the opinion of the investigator would impact the study outcomes.
13. If taking chronic medications (e.g., anti-hypertensive medications), they must have been taking the product for at least two months to screening and agree to maintain the same dosage throughout the study.
14. Has severe or uncontrolled type 2 diabetes, psychiatric disorder, gastrointestinal disease (i.e., diarrhoea, Crohn's disease, ulcerative colitis, IBS, diverticulosis, stomach or duodenal ulcers respiratory or cardiac illness or any other condition which in the opinion of the investigator would impact the study outcomes.
15. Has a current or history of any gastrointestinal cancer
16. Are severely immunocompromised (HIV positive, transplant patient, on anti-rejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy with the last year).
17. Experiences alarm features such as weight loss, rectal bleeding, a recent change in bowel habit (<3 months).
18. Have a current malignant disease or any concomitant end-stage organ disease.
19. Individuals who, in the opinion of the investigator are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
20. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.
21. Participants who have undergone intensive skin treatments (e.g. laser treatment or skin related surgery) in the last 3 months.
22. If taking any dietary supplements or medications known to affect skin health or other trial measures (resveratrol, ginkgo biloba, ginseng, fruit powder extracts and DHA).
23. Has a skin condition likely to interfere with skin assessments (e.g., eczema, dermatitis, any open skin wounds, reactive and sensitive skin).

    -

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Faecal microbial composition and diversity | from baseline to 12 weeks
  To assess the changes of faecal microbial composition and diversity from baseline to 12 weeks supplementation of three different doses of colon delivered vitamin B2 to compare the changes to placebo. levels, and alpha and beta diversity indices at the genus and species level as measured by metagenomic based profiles at baseline and at week 12

SECONDARY OUTCOMES:
Faecal microbial metabolites fatty acid content at baseline and week 12 | Intestinal inflammation as assessed by faecal calprotectin at baseline and at week 12
  Faecal microbial metabolites measured as short-chain fatty acid content at baseline and week 12
Intestinal inflammation | from baseline to 12 weeks
  Intestinal barrier integrity as assessed by sCD14 at baseline and at week 12
Intestinal barrier integrity | from baseline to 12 weeks
  Oxidative stress level measured as free thiol content in blood at baseline and at week 12
Oxidative stress in blood | from baseline to 12 weeks
  Oxidative stress level measured as free thiol content in blood at baseline and at week 12
Inflammatory status in blood | from baseline to 12 weeks
  Systemic inflammation measured as high sensitive C reactive protein (hs-CRP) in blood at baseline and at week 12.
Gastrointestinal symptoms | from baseline to 12 weeks
  Gastrointestinal symptoms as assessed by Gastrointestinal Symptom Rating Scale (GSRS).The GSRS is a 15 items questionnaire combined into five symptom clusters i.e Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.(GSRS) at baseline and at week 12.
health-related quality of life | from baseline to 12 weeks
  Quality of life as assessed by short form survey-36 (SF-36) questionnaires at baseline and at week 12.
  The SF-36 is a self-administered questionnaire comprising 36-items measuring eight health domains: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). These outcomes will be grouped as a physical component summary and a mental component summary. The norm data is 0-100, and the health-related quality of life increases as the scores increase.
Stool consistency | from baseline to 12 weeks
  Stool consistency (Bristol Stool Scale), as reported in the daily eDiary app (at baseline and week 12).
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). 'Normal' stool is considered to be Types 3 and 4; and Types 6 and 7 would be considered to suggest mild and severe diarrhea, respectively.
Stool frequency | from baseline to 12 weeks
  Stool frequency, as reported in the daily eDiary app (at baseline and week 12).
Systemic vitamin status | from baseline to 12 weeks
  The concentration of B vitamins in blood at baseline
Faecal physiological pH | from baseline to 12 weeks
  Faecal physiological parameters measured as pH potential at baseline and at week 12.
Faecal microbial composition and diversity at week 4 | from baseline to 4 weeks
  Faecal microbial composition at phylum, genus, and species levels, and alpha and beta diversity indices at the genus and species level as measured by metagenomic based profiles at baseline and at week 4.
Microbial metabolites at week 4 | from baseline to 4 weeks
  Faecal microbial metabolites measured as short-chain fatty acid content at baseline and week 4.

OTHER OUTCOMES:
Skin barrier integrity | from baseline to 12 weeks
  Skin barrier integrity measured as trans-epidermal water loss (TEWL) g/m²/h at baseline and at week 12.
Skin hydration | from baseline to 12 weeks
  Skin hydration measured using corneometry from 0 (no water at all) to 120 (on water) at baseline and at week 12.
Objective skin-health | from baseline to 12 weeks
  Objective skin-health assessment completed by the participant using Likert scale (from not at al to very much) at baseline and at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Timothy Dinan, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical Trials, 1st Floor, Block C, Heron House, Blackpool Retail Park, Cork, Cork, Ireland